CLINICAL TRIAL: NCT01707784
Title: Effects of Stress on Glucose Tolerance During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Jardena Puder, MD, University of Lausanne Hospitals
Other Study IDs: 295/12
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy; Stress; Gestational Diabetes
Keywords: Pregnancy; Stress; Anxiety; Cortisol; Copeptin; Gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational; Anxiety Disorders; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with gestational diabetes: Women with gestational diabetes diagnosed by clinically routine 75 g oral glucose tolerance testing
- Women without gestational diabetes: Women without gestational diabetes diagnosed by clinically routine 75 g oral glucose tolerance testing

SUMMARY:
The objective of the study is to investigate the effect of stress on glucose tolerance during pregnancy.

The main objectives of the study are to investigate if various measures of stress (stressful life events, the perceived level of stress and the cortisol or copeptin concentrations) differ between pregnant women with and without gestational diabetes during the end of the second/beginning of the third trimester when presenting for their routine glucose tolerance testing.

Secondary objectives are the link between these different stress measures and the routinely measured fasting and stimulated glucose levels during the oral glucose tolerance test.

DETAILED DESCRIPTION:
Hypotheses in this study, 3 primary hypotheses will be tested.

1. Women with gestational diabetes have more life events compared to pregnant women without gestational diabetes.
2. Women with gestational diabetes have higher perceived level of stress and anxiety compared to pregnant women without gestational diabetes.
3. Women with gestational diabetes have higher measures of cortisol levels in the saliva and in the nailfolds and higher plasma copeptin levels compared to pregnant women without gestational diabetes.

Secondary objectives:

1. To test the link between these stress measures and the fasting and stimulated glucose levels during the oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who are undergoing a 75 g oral glucose tolerance test at the "Maternité" of CHUV at 24-30 weeks of gestation between October 2012 and April 2013

Exclusion Criteria:

* Pregnant woman who has the use if medications that influence either the cortisol and /or the glucose levels
* Pregnant woman who has the inability to fill out the questionnaires with assistance

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Markers of stress | At assessment
  stress (stressful life events, the perceived level of stress and the cortisol or copeptin concentrations)

CONTACTS AND LOCATIONS:
Overall Officials: Jardena J. Puder, MD, Study Director — University of Lausanne; Ji-Seon Kang, Principal Investigator — University of Lausanne; Yvan Vial, MD, Principal Investigator — University of Lausanne; Pr Ulrike Ehlert, PhD, Principal Investigator — University of Zurich; Ayala Borghini, PhD, Principal Investigator — University of Lausanne; Pedro Marques-Vidal, MD, PhD, Principal Investigator — University of Lausanne
Locations (1):
- Maternité CHUV, University of Lausanne, Lausanne, Switzerland